CLINICAL TRIAL: NCT03398213
Title: Acupuncture Efficacy in the Treatment of Acute Exacerbations of Chronic Obstructive Pulmonary Disease During Hospitalization: a Randomized Controlled Trial
Brief Title: Acupuncture Treatment of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0108-17-BNZ
Record Dates: First submitted 2017-12-31; First posted 2018-01-12 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2019-06

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental): Acupuncture for treatment of COPD exacerbation + standard conventional care for COPD exacerbation
  Interventions: Other: Acupuncture
- Sham procedure (Sham Comparator): Ear stimulation with plaster + standard conventional care for COPD exacerbation
  Interventions: Other: Sham procedure
- Standard care (No Intervention): Standard conventional care for COPD exacerbation

INTERVENTIONS:
Other: Acupuncture — Acupuncture
  Arms: Acupuncture
Other: Sham procedure — Ear stimulation with plaster
  Arms: Sham procedure

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major health problem. Acute exacerbations are a health-care burden involving frequent hospitalizations and elevated costs. They have effective therapies with significant side effects. Acupuncture has been shown to reduce dyspnea and other COPD-related symptoms. The investigators will compare the efficacy and safety of the addition of true acupuncture to usual care with both sham-acupressure added to usual care and usual care only for the treatment of acute exacerbations of COPD among inpatients.

DETAILED DESCRIPTION:
This is an assessor-blinded randomized controlled trial in the setting of a tertiary academic medical center in Israel. Patients with clinical diagnosis of acute exacerbation of COPD will be randomized to either usual care only, usual care with true acupuncture or usual care with sham-acupressure. The primary outcome will be clinical improvement of dyspnea as measured by mBorg scale. Secondary outcomes included improvement of other patient-reported outcomes and physiologic features, as well as duration of hospitalization and treatment failure. Acupuncture-related side effects will be evaluated by the validated Acupuncture Adverse Events (AcupAE) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of COPD
* Clinical diagnosis of acute exacerbation of COPD
* Informed consent

Exclusion Criteria:

* Hemodynamic instability
* Platelet count < 20 x 10^9/L
* Expected respiratory deterioration requiring mechanical ventilation in the next 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, M.D., Principal Investigator — Bnai Zion Medical Center
Locations (2):
- Israel (2):
  - Bnai Zion Medical Center, Haifa, Golomb 47
  - Bnai Zion Medical Center, Haifa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy I, Elimeleh Y, Gavrieli S, Attias S, Schiff A, Oliven A, Schiff E. Treatment of acute exacerbations of chronic obstructive pulmonary disease with acupuncture during hospitalization: a three-arm double-blinded randomized sham-controlled trial. Acupunct Med. 2022 Dec;40(6):505-515. doi: 10.1177/09645284221086293. Epub 2022 May 17. PMID 35579025

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture: Acupuncture for treatment of COPD exacerbation + standard conventional care for COPD exacerbation
  Acupuncture: Acupuncture
  N=26
- Sham Procedure: Ear stimulation with plaster + standard conventional care for COPD exacerbation
  Sham procedure: Ear stimulation with plaster
  N=24
- Standard Care: Standard conventional care for COPD exacerbation
  N=22
Period: Overall Study
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Started | 26 | 24 | 22
Completed | 26 | 24 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Procedure | Standard Care | Total
Number analyzed (Participants) | 26 | 24 | 22 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (10.1) | 70.7 (8.1) | 67.4 (9.3) | 69.13 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 5 | 20
  Male | 20 | 15 | 17 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Dyspnea intensity [Median (Inter-Quartile Range); unit: units on a scale] | 8 [5.5 to 8.75] | 6.5 [5 to 8.5] | 7.75 [6 to 8.5] | 7.5 [5 to 8.5]

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea Intensity
Description: modified Borg (mBorg) scale, which is a validated scale that has been used to evaluate the degree of dyspnea (0- no dyspnea, to 10- worse dyspnea)
Time Frame: At baseline, day 1 after treatment, day 2 before treatment, day 2 after treatment, day 3 before treatment, day 3 after treatment, day 4 before treatment, and day 4 after treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
units on a scale
  Baseline | 8.0 [5.5 to 8.75] | 6.5 [5.0 to 8.5] | 7.75 [6.0 to 8.5]
  Day 1 after treatment | 5 [4.0 to 5.0] | 6 [4.25 to 7.8] | 7 [5.5 to 8.0]
  Day 2 before treatment | 5 [3.5 to 7] | 6.75 [5 to 8.5] | 7.5 [5.8 to 8.3]
  Day 2 after treatment | 2 [1 to 3] | 5 [3 to 7] | 7.5 [5 to 8]
  Day 3 before treatment | 2.5 [1 to 5] | 6 [4.5 to 7.3] | 5.75 [4.5 to 7]
  Day 3 after treatment | 2 [1 to 3] | 6 [5 to 7] | 6 [2 to 7]
  Day 4 before treatment | 3 [0 to 5] | 5.5 [3 to 8] | 7 [5 to 8.5]
  Day 4 after treatment | 1 [0 to 3] | 5 [4 to 6] | 6 [5 to 7]

2. Secondary Outcome: Duration of Hospitalization
Description: Days of hospitalization
Time Frame: Through study completion, an average of 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
days | 5.5 (2.3) | 6.0 (2.9) | 6.3 (2.9)

3. Secondary Outcome: Carbon Dioxide Partial Pressure (pCO2)
Description: pCO2
Time Frame: Day 1, day 2, day 3, and day 4 of the study
Population: Blood gases were not taken daily to all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
Participants
  Day 1: < 45 mmHg | 6 | 3 | 8
  Day 1: 45-60 mmHg | 12 | 17 | 9
  Day 1: 60-80 mmHg | 5 | 4 | 5
  Day 1: > 80 mmHg | 3 | 0 | 0
  Day 2: number analyzed (Participants) | 18 | 19 | 8
  Day 2: < 45 mmHg | 4 | 7 | 1
  Day 2: 45-60 mmHg | 4 | 6 | 3
  Day 2: 60-80 mmHg | 7 | 5 | 2
  Day 2: > 80 mmHg | 3 | 1 | 2
  Day 3: number analyzed (Participants) | 12 | 15 | 9
  Day 3: < 45 mmHg | 1 | 3 | 4
  Day 3: 45-60 mmHg | 5 | 9 | 3
  Day 3: 60-80 mmHg | 4 | 2 | 1
  Day 3: > 80 mmHg | 2 | 1 | 1
  Day 4: number analyzed (Participants) | 6 | 11 | 6
  Day 4: < 45 mmHg | 1 | 2 | 2
  Day 4: 45-60 mmHg | 1 | 6 | 0
  Day 4: 60-80 mmHg | 3 | 3 | 3
  Day 4: > 80 mmHg | 1 | 0 | 1

4. Secondary Outcome: Power of Hydrogen (pH)
Description: pH
Time Frame: Day 1, day 2, day 3, and day 4 of the study
Population: Blood gases were not measured daily in all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
Participants
  Day 1: < 7.2 | 0 | 0 | 0
  Day 1: 7.2-7.3 | 5 | 4 | 1
  Day 1: > 7.3 | 21 | 20 | 21
  Day 2: number analyzed (Participants) | 18 | 19 | 8
  Day 2: < 7.2 | 0 | 0 | 0
  Day 2: 7.2-7.3 | 6 | 3 | 4
  Day 2: > 7.3 | 12 | 16 | 4
  Day 3: number analyzed (Participants) | 9 | 15 | 9
  Day 3: < 7.2 | 0 | 1 | 0
  Day 3: 7.2-7.3 | 2 | 0 | 2
  Day 3: > 7.3 | 7 | 14 | 7
  Day 4: number analyzed (Participants) | 6 | 11 | 6
  Day 4: < 7.2 | 0 | 0 | 0
  Day 4: 7.2-7.3 | 0 | 0 | 2
  Day 4: > 7.3 | 6 | 11 | 4

5. Secondary Outcome: Respiratory Rate
Description: Respiratory rate
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: breaths per minute
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
breaths per minute
  Baseline (day 1) | 21 [16 to 23.75] | 22 [16.5 to 26] | 20 [16 to 22]
  Day 1 after treatment | 16 [14 to 20] | 18 [16 to 20.5] | 21 [18 to 26]
  Day 2 before treatment | 18 [16 to 22] | 20 [16 to 25] | 22 [16 to 24]
  Day 2 after treatment | 16 [12 to 16] | 18 [16 to 21.5] | 26 [21 to 30]
  Day 3 before treatment | 16 [14 to 29] | 18 [16 to 24] | 18 [16 to 22]
  Day 3 after treatment | 14 [12 to 20] | 16 [16 to 24] | 24 [18 to 24]
  Day 4 before treatment | 16 [14 to 29] | 16 [16 to 23] | 18 [16 to 18]
  Day 4 after treatment | 13 [12 to 17] | 16 [14 to 20] | 22 [18 to 26]

6. Secondary Outcome: Oxygen Saturation
Description: Oxygen saturation
Time Frame: Day 1, day 2, day 3, and day 4 of the study
Population: Oxygen saturation is missing for some participants in days 2, 3 and 4
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
Participants
  Day 1: =< 80% | 4 | 1 | 0
  Day 1: 81-89% | 9 | 10 | 10
  Day 1: >= 90% | 13 | 13 | 12
  Day 2: number analyzed (Participants) | 24 | 24 | 19
  Day 2: =< 80% | 2 | 4 | 2
  Day 2: 81-89% | 10 | 10 | 5
  Day 2: >= 90% | 12 | 10 | 12
  Day 3: number analyzed (Participants) | 19 | 23 | 17
  Day 3: =< 80% | 0 | 3 | 0
  Day 3: 81-89% | 10 | 7 | 6
  Day 3: >= 90% | 9 | 13 | 11
  Day 4: number analyzed (Participants) | 11 | 17 | 14
  Day 4: =< 80% | 1 | 0 | 0
  Day 4: 81-89% | 4 | 3 | 2
  Day 4: >= 90% | 6 | 14 | 12

7. Secondary Outcome: Cough Intensity
Description: Visual Analogue Scale (VAS) for cough (0- no cough, to 10- worse cough)
Time Frame: Day 1, day 2, day 3, and day 4 of the study
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
units on a scale
  Day 1 | 7.5 [5.0 to 8.0] | 5.0 [5.0 to 7.3] | 5.0 [4 to 7.5]
  Day 2 | 4.5 [1.5 to 5.5] | 5 [2.5 to 7.5] | 5 [4.5 to 7.5]
  Day 3 | 3 [1 to 5] | 5 [3.3 to 7.3] | 5 [2.5 to 7.5]
  Day 4 | 2.5 [2 to 4] | 4.5 [2.5 to 6] | 5 [0 to 7.5]

8. Secondary Outcome: Sputum Intensity
Description: Visual Analogue Scale (VAS) for sputum (0- no sputum, to 10- worse sputum)
Time Frame: Day 1, day 2, day 3, and day 4 of the study
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acupuncture | Sham Procedure | Standard Care
Number analyzed (Participants) | 26 | 24 | 22
units on a scale
  Day 1 | 6.0 [2 to 7.5] | 6.0 [4.5 to 6.0] | 5.0 [2.5 to 6.0]
  Day 2 | 2.8 [1 to 4.5] | 5.5 [2 to 6] | 4.5 [2.5 to 5.5]
  Day 3 | 2 [1 to 4] | 5 [3.5 to 6] | 4.5 [2.5 to 5]
  Day 4 | 2 [1 to 4] | 5 [3 to 6] | 5 [2.5 to 6]

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Acupuncture | Sham Procedure | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03398213/Prot_SAP_000.pdf